CLINICAL TRIAL: NCT06771063
Title: A Multicenter, Randomized, Double-blind, Positive-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of WXSH0102 Tablets in the Treatment of Vulvovaginal Candidiasis (VVC)
Brief Title: A Study of the Efficacy and Safety of WXSH0102 in Treating VCC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cisen Pharmaceutical CO., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WXSH0102-02-001
Record Dates: First submitted 2024-12-25; First posted 2025-01-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Vaginitis
MeSH Terms: conditions — Vaginitis | interventions — Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A : WXSH0102 Day1 1400 mg Day2-3 700 (Experimental): Arm A will receive WXSH0102 tablets with a loading dose of 1400 mg on the first day followed by a maintenance dose of 700 mg for two consecutive days
  Interventions: Drug: WXSH0102/placebo
- Arm B : WXSH0102 Day1 1000 mg Day2-3 500 arm (Experimental): Arm B will receive WXSH0102 tablets with a loading dose of 1000 mg on the first day followed by a maintenance dose of 500 mg for two consecutive days
  Interventions: Drug: WXSH0102/placebo
- C : WXSH0102 Day1 600 mg Day2-3 300 (Experimental): Arm C will receive WXSH0102 tablets with a loading dose of 600 mg on the first day followed by a maintenance dose of 300 mg for two consecutive days
  Interventions: Drug: WXSH0102/placebo
- Arm D: fluconazole (Active Comparator): Arm D (active control group) will receive fluconazole capsules for only one day on D1
  Interventions: Drug: fluconazole capsules/placebo

INTERVENTIONS:
Drug: WXSH0102/placebo — Administer WXSH0102 tablets/placebo orally.
  Arms: Arm A : WXSH0102 Day1 1400 mg Day2-3 700; Arm B : WXSH0102 Day1 1000 mg Day2-3 500 arm; C : WXSH0102 Day1 600 mg Day2-3 300
Drug: fluconazole capsules/placebo — Administer fluconazole capsules/placebo orally
  Arms: Arm D: fluconazole

SUMMARY:
This study is a multicenter, randomized, double-blind, active-controlled, dose-ranging clinical trial designed to evaluate the efficacy and safety of the investigational drug compared to the active comparator in the treatment of vulvovaginal candidiasis. The trial consists of three phases: screening/enrollment (D-3 to D-1), treatment period (D1 to D3), and follow-up period (D4, D11±2, D25±3). Eligible subjects in this study will be randomized in a 1:1:1:1 ratio to three investigational drug arms with different dosing regimens and one active control arm. Specifically, Group A will receive WXSH0102 tablets with 1400 mg on the first day followed by a maintenance dose of 700 mg for two consecutive days, Group B will receive WXSH0102 tablets with 1000 mg on the first day followed by a maintenance dose of 500 mg for two consecutive days, Group C will receive WXSH0102 tablets with 600 mg on the first day followed by a maintenance dose of 300 mg for two consecutive days, and Group D (active control group) will receive fluconazole capsules for only one day on D1. All medications will be administered orally.

ELIGIBILITY:
Inclusion Criteria:

* The subjects understood and voluntarily signed the informed consent Form (ICF), and were willing and able to comply with the study protocol.
* Female participants who signed ICF at the age of 18-64 years (including the cut-off value) and had sexual intercourse;
* Participants were diagnosed with VVC and met each of the following criteria: a. At screening, the total score on the VVC scale was ≥4 and at least two of the symptoms or signs on the VVC scale were present; b. A vaginal discharge sample collected at screening was Gram stain positive for Candida (hypha/pseudohypha/budding); c. Vaginal pH ≤4.5; Symptoms: vulvovaginal itching, vulvar burning pain, dyspareunia and urination pain, excessive secretion, secretion is tofu residue like; Physical signs: gynecological examination showed vulvar hyperemia and edema, which may be accompanied by scratches. In severe cases, chapped skin, exfoliation and even erosion could be seen. Vaginal mucosa was hyperemic, vaginal secretion was curd or tofu residue like;
* Subjects who are capable of oral administration;
* For the duration of the study, participants agreed to abstain from sexual activity and to use the condom throughout sexual activity.

Exclusion Criteria:

* Known or suspected allergic history to any component of this product, fluconazole or pyrrole drugs;
* Subjects with any vulvovaginal or cervical disease that may affect the diagnosis and evaluation of VVC;
* Topical or systemic antifungal treatment for VVC within 14 days before randomization;
* Significant liver disease or abnormal liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST] > 1.5 ULN); Patients with severe renal disease or renal insufficiency (glomerular filtration rate (GFR) < 60ml/min/1.73m2 );
* Patients who planned to undergo treatment or surgery for vulvar, vaginal or cervical lesions during the study period;
* Severe gastrointestinal disease or other conditions that may affect the absorption of the trial drug;
* Patients with severe heart, lung, liver, kidney dysfunction and hematopoietic system diseases;

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 108 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving cure at the D11±2 visit. | day 11±2
  Proportion of subjects achieving cure (defined as the disappearance of VVC symptoms and signs along with a negative Candida culture) at the D11±2 visit.

SECONDARY OUTCOMES:
Proportion of subjects achieving clinical cure at the D11±2 visit | day 11±2
  Proportion of subjects achieving clinical cure (complete disappearance of VVC symptoms and signs) at the D11±2 visit;
Proportion of subjects achieving mycological clearance at the D11±2 visit | day 11±2
  Proportion of subjects achieving mycological clearance (negative growth of Candida species in fungal culture) at the D11±2 visit;
Proportion of subjects achieving clinical improvement at the D11±2 visit | day 11±2
  Proportion of subjects achieving clinical improvement (partial or complete resolution of symptoms and signs, with a total VVC scale score ≤1) at the D11±2 visit
Difference in VVC scale scores between the D11±2 visit and baseline visit | day 11±2
  Difference in VVC scale scores between the D11±2 visit and baseline visit
Proportion of subjects achieving cure at the D25±3 visit. | Day 25±3
  Proportion of subjects achieving cure (defined as the disappearance of VVC symptoms and signs along with a negative Candida culture) at the D25±3 visit..
Proportion of subjects achieving mycological clearance at the D25±3 visit | Day 25±3
  Description: Proportion of subjects achieving mycological clearance (negative growth of Candida species in fungal culture) at the D25±3 visit;
Proportion of subjects achieving clinical improvement at the D25±3 visit | Day 25±3
  Description: Proportion of subjects achieving clinical improvement (partial or complete resolution of symptoms and signs, with a total VVC scale score ≤1) at the D25±3visit
Proportion of subjects requiring rescue therapy during the trial; | Day 25±3
  Proportion of subjects requiring rescue therapy during the trial;
Proportion of subjects with normal vaginal microecology assessments | Day11±2 and day 25±3
  Proportion of subjects with normal vaginal microecology assessments at the D11±2 and D25±3 visits
adverse events | Day 25±3
  Incidence and severity of adverse events and serious adverse events
AUC0-tau | day 4
  the AUC0-tau estimated using non-compartmental and/or population pharmacokinetic models
Cmax | day 4
  the Cmax estimated using non-compartmental and/or population pharmacokinetic models

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - 251 Yaojiayuan Road, Chaoyang District, Beijing, Beijing, Beijing Municipality
  - Beijing Obstetrics and Gynecology Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided